CLINICAL TRIAL: NCT02679820
Title: PostPlacental IUD Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Lecturer of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LA010516
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PostPlacental IUD insertion (Experimental): Copper T intrauterine device will be inserted immediately following delivery of the placenta in cases of cesarean section deliveries.
  Interventions: Device: Copper T intrauterine device
- Control (No Intervention): IUD will be offered as a method of contraception after puerperium

INTERVENTIONS:
Device: Copper T intrauterine device
  Other Names: copper T IUD
  Arms: PostPlacental IUD insertion

SUMMARY:
The immediate post cesarean section IUD insertion is a further step towards spreading more compliance to females in developing countries, with rapid increase in population size

ELIGIBILITY:
Inclusion Criteria:

* Females desiring contraception by using intrauterine device following their vaginal delivery or cesarean section

Exclusion Criteria:

* refusal to participate in the study
* desiring other methods of contraception
* will not use any method of contraception
* has a contraindication for the use of IUD as bicornuate or septate uterus, sub mucous myomas, etc.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Expulsion rate | 6 months
The percentage of females seeking contraception | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina MR Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bayoumi YA, Dakhly DMR, Bassiouny YA, Gouda HM, Hassan MA, Hassan AA. Post-placental intrauterine device insertion vs puerperal insertion in women undergoing caesarean delivery in Egypt: a 1 year randomised controlled trial. Eur J Contracept Reprod Health Care. 2020 Dec;25(6):439-444. doi: 10.1080/13625187.2020.1823366. Epub 2020 Oct 2. PMID 33006501